CLINICAL TRIAL: NCT06568861
Title: A Phase 1 Non-Randomized, Open-Label, Multiple Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ALG-097558 in Subjects With Moderate Hepatic Impairment and in Healthy Subjects With Normal Hepatic Function
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ALG-097558 in Subjects With Hepatic Impairment and in Healthy Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALG-097558-702 / DMID 24-0001
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study is non-randomized, open-label, parallel group study. Cohort 1 will enroll moderately hepatically impaired subjects and Cohort 2 will enroll subjects without hepatic impairment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with Moderate Hepatic Impairment (Child-Pughs Class B) (Experimental): Subjects with moderate hepatic impairment will receive oral doses of 200 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558
- Subjects with Normal Hepatic Function (Experimental): Subjects with normal hepatic function will receive oral doses of 200 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558

INTERVENTIONS:
Drug: ALG-097558 — Multiple doses of ALG-097558 200 mg (2 x 100 mg tablets)

SUMMARY:
This is a Phase 1 non-randomized, open-label, multiple dose, parallel-group study of ALG-097558 in subjects with moderate hepatic impairment and subjects without hepatic impairment, matched for age, body weight and, to the extent possible, for gender. The primary purpose of this study is to characterize the effect of hepatic impairment on the plasma pharmacokinetics of ALG-097558 following administration of multiple, twice daily (Q12H) oral (PO) doses.

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Male and Female between 18 and 75 years old
2. BMI 17.5 to 40.0 kg/m^2 and a total body weight >50 kg (110 lb) 3 .Female subjects must either be not of childbearing potential or if they are a woman of childbearing potential, they are only eligible if they and any non-sterile, male sexual partners agree to use highly effective contraceptive therapy

4. Female subjects must have a negative serum pregnancy test at screening

Inclusion Criteria for Subjects with Normal Hepatic Function:

1. Good general health as defined by no clinically relevant abnormalities identified by Medical History and a vital signs and 12-lead electrocardiogram (ECG) assessment
2. Subjects must fit the demographic-matching criteria including body weight, age, and to the extent possible, gender
3. Normal hepatic function with no known or suspected hepatic impairment

Inclusion Criteria for Subjects with Impaired Hepatic Function:

1. Subject satisfies the criteria for Class B of the Child-Pugh classification (Child Pugh Scores 7-9 points) within 28 days of study drug administration
2. A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination, liver biopsy, hepatic ultrasound, Fibroscan, computerized tomography scan, or magnetic resonance imaging (MRI)
3. Stable hepatic impairment for at least 3 months prior to screening or second screening visit to demonstrate stability
4. Stable concomitant medications for the management of an individual subject's medical history for at least 28 days prior to screening
5. Subjects must have a 12-lead ECG and vital signs assessment that meet the protocol criteria

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subjects with a recent (within 1 year of randomization) history or current evidence of drug abuse or recreational drug use
5. Excessive use of alcohol defined as regular consumption of ≥14 units/ week for women and ≥21 units/week for men
6. Unwilling to abstain from alcohol use for 48 hours prior to start of the study through end of study follow up
7. Subjects with Hepatitis A, B, C, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection. Subejcts with Hepatitis B infection may be eligible for moderate impairment cohort provided provided they met stable treatment criteria. Subjects with HIV infection may be eligible for moderate impairment cohort provided they met stable treatment criteria.

Exclusion Criteria for Subjects with Normal Hepatic Function:

1. Estimated creatinine clearance <60 mL/min/1.73 m2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula] - Unless otherwise instructed by the Study Review Committee (SRC), CKD-EPI should not be corrected for subjects of African ancestry
2. Bilirubin (total, direct) >1.2× upper limit of normal (ULN) (unless Gilbert's is suspected)
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > 1.2×ULN
4. Grade ≥1 Hemoglobin

Exclusion Criteria for Subjects with Impaired Hepatic Function:

1. Subjects with advanced ascites (Grade 3)
2. Subjects with refractory encephalopathy as judged by the investigator.
3. Subjects with esophageal variceal bleeding within the past 6 months prior to screening.
4. Subjects with Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement.
5. Estimated creatinine clearance <60 mL/min/1.73 m2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula] - Unless otherwise instructed by the SRC, CKD-EPI should not be corrected for subjects of African ancestry
6. ALT or AST level ≥5×ULN
7. Serum sodium ≤125 mmol/L
8. Platelets <50×10^9/L
9. Grade ≥2 Hemoglobin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma
Time to maximum plasma concentration [Tmax] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma
Maximum plasma concentration [Cmax] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma
Minimum plasma concentration [Cmin] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma
C0 [predose] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma
Half-life [t1/2] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 in plasma

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 20 Days
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida